CLINICAL TRIAL: NCT06805994
Title: Parent-to-Child Nasal Microbiota Transplant to Reestablish Nasal Microbiome Diversity After Intranasal Mupirocin Treatment of Children With Staphylococcus Aureus Nasal Colonization
Brief Title: Administering NMT to Reestablish Infant Nasal Microbiome Diversity Following Intranasal Mupirocin Treatment
Acronym: NMT Protocol 3
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00480834
Record Dates: First submitted 2025-01-28; First posted 2025-02-03 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Staphylococcal Aureus Infection; Microbial Colonization; Pediatric Infection; S. Aureus Colonization; Microbial Transplant
Keywords: microbiome; s. aureus; staph
MeSH Terms: conditions — Communicable Diseases; Staphylococcal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Single NMT (Experimental): Swab parent nares then insert swab directly into child nares once.
  Interventions: Biological: Nasal Microbiota Transplant (NMT)
- Repeat NMT (Experimental): Swab parents nares then insert swab directly into child nares multiple times.
  Interventions: Biological: Nasal Microbiota Transplant (NMT)
- Placebo (Placebo Comparator): Insert a sterile swab into child nares.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Nasal Microbiota Transplant (NMT) — nasal microbiota transplant
  Arms: Repeat NMT; Single NMT
Biological: Placebo — Placebo sterile swab
  Arms: Placebo

SUMMARY:
This protocol aims to evaluate how NMT affects pediatric nasal microbiome diversity following intranasal mupirocin treatment

DETAILED DESCRIPTION:
This parent-to-child NMT study will test the effect of an anterior nares, or nasal, microbiota transplant (NMT) on seeding, engraftment, and diversity of the neonatal microbiome following nasal decolonization for S. aureus. Infants admitted to the Johns Hopkins Neonatal Intensive Care Unit (NICU) will be screened and parents will be approached for enrollment in the study. After consent and baseline screening of parents and infants, eligible infants will undergo an NMT.

ELIGIBILITY:
Child:

Inclusion criteria

1. Child has had a prior nasal surveillance culture grow S. aurues
2. Child is <18 years of age
3. Child completed treatment with intranasal mupirocin for S. aureus nasal colonization as part of routine clinical care two or more days before the planned transplant
4. Child has anticipated hospital length of stay >3 days after completing intranasal mupirocin treatment
5. Infant >25 weeks gestation unless >2 months chronological age

Exclusion criteria

1. Child is a ward of the State
2. Child with a diagnosis of immunodeficiency or antenatal suspicion for immunodeficiency (e.g., sibling with known immunodeficiency, genetic syndrome with known associated immunodeficiency)
3. Child cannot have nasal swabs collected (due to anatomic or other clinical intervention, including nasal packing)

Donor:

Inclusion criteria

1. Donor is able to provide informed consent
2. Donor has a relationship with the child outside of the hospital setting (i.e., not an ICU caregiver)

Exclusion criteria

1. Donor had positive COVID-19 test in prior 21 days
2. Donor with signs or symptoms of respiratory illness (e.g. runny nose, congestion, fever, cough)
3. Donor has been in close contact with someone in the last 7 days who had a respiratory viral infection (e.g., cold, flu)
4. Donor tests positive on baseline screening test for S. aureus nasal colonization.
5. Donor tests positive on baseline screening test for a respiratory pathogen.
6. Donor is not able to provide written informed consent
7. Donor is not able to be present at the bedside at the time of intervention.
8. Donor has history of chronic sinusitis, cystic fibrosis, or an infection with a multi-drug resistant organism.
9. Inability or unwillingness to complete the Donor questionnaire or a positive response to any question on the Donor questionnaire.
10. Donor has smoked within the last month

Ages: 0 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 175 (Estimated)
Dates: Start 2025-08-27 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Pediatric nasal microbiome diversity after parent-to-child NMT. | Day 2, 4, 7, 10, 14 days post-intervention
  This outcome will be determined by analysis of periodic surveillance swabs collected after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron M Milstone, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No